CLINICAL TRIAL: NCT02679482
Title: Following Patients After Selective and Pascal Laser Trabeculoplasty for Treatment of Chronic Open-Angle Glaucoma
Acronym: FPSPLTTCOAG
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fundación Oftalmológica Nacional (Other)
Responsible Party: Sponsor
Other Study IDs: FONCI6001
Record Dates: First submitted 2016-02-06; First posted 2016-02-10 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-02

CONDITIONS: Glaucoma, Open-Angle; Glaucoma, Primary Open Angle; Exfoliation Glaucoma; Glaucoma, Pigmentary
Keywords: Primary Open Angle Glaucoma; Selective Laser Trabeculoplasty; Pattern Scan Laser Trabeculoplasty
MeSH Terms: conditions — Glaucoma, Open-Angle; Exfoliation Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Selective laser trabeculoplasty (SLT): Patients who underwent to Selective laser trabeculoplasty
- Pattern laser trabeculoplasty (PLT): Patients who underwent to Pattern laser trabeculoplasty

SUMMARY:
The purpose of this study is to follow and describe the outcomes of patients after selective and pascal laser trabeculoplasty treatment for chronic open-angle glaucoma.

DETAILED DESCRIPTION:
Selective laser trabeculoplasty (SLT) and pattern laser trabeculoplasty (PLT, a novel computer-guided laser that is being using to treat open-angle glaucoma) are two laser surgery methods to make a trabeculoplasty on patients with open angle glaucoma. An observational prospective study will be performed, a consecutive convenience sample patients with indication for SLT or PLT will be recruited during June 2014 to uly 2016 and follow-up until 6 months, at the Fundación Oftalmológica Nacional (Bogotá-Colombia). A non-probabilistic convenience sampling is performed, considering that the average number of patients diagnosed with chronic open-angle glaucoma undergoing to Laser trabeculoplasty at the Oftalmológica Nacional Fundacion corresponds to approximate 2 per month. Therefore it is expected to enroll one patient per month for each of the laser used (SLT and PLT) for trabeculoplasty. Finally obtaining a sample size of 18 patients per type of laser for a total of 36 patients in the recruitment period, between September 2014 and July 2016.

This study is strictly observational, that's why the laser procedure is covered by the national health insurance of each patient, as well the complications due to the same procedure. An evaluation pre trabeculoplasty and a consecutive 5 visits will be perform as follows:

Visit 0 - Pre-procedure visit: the subjects that will undergo laser trabeculoplasty either Selective laser or PASCAL laser will be invited to participate and an informed consent will be carried out. The information concerting to demographics characteristics (study eye, age, gender and ethnicity), clinical characteristics (date of glaucoma diagnosis, number of medications used to treat glaucoma, time of use of actually anti-glaucomatous topical medication) and slit lamp and ophthalmoscopy examination (corneal aspect, iris color, pupil gonioscopy, intraocular pressure, lens status, vitreous cells, vertical C/D ratio, optic nerve edge, rim characteristic [ISNT pattern], peripapilar atrophy, state of fovea, state of peripheral retina and state of choroid for both eyes) will be extracted and recorded on respective case report form (CRF). The data will be scored according to the grading criteria outlined below:

Study eye: the eye under the follow-up 0 - Right eye 1 - Left eye

Geder: the state of being male or female 0 - Male 1 - Female

Ethnicity: the fact or state of belonging to a social group that has a common national or cultural tradition.

0 - Hispanic

1. - Black
2. - White
3. - Asian

Number of medications used: anti-glaucoma medication used by the patient 0 - 0

1. - 1
2. - 2
3. - 3
4. - 4

Corneal aspect: state in which the cornea is at baseline 0 - Normal 1 - Anormal

Iris color: iris pigmentation 0 - Light

1. - Medium
2. - Dark

Gonioscopy (Shaffer classification): amplitude of irido-corneal angle maseure by poster lens and noted by the Shaffer scale on each quadrant superior, nasal, temporal and inferor angle 0 - 0

1. - 1
2. - 2
3. - 3
4. - 4

Intraocular pressure: pressure inside the eye measured in millimeters of mercury Value in mmhg, measure with Goldman tonometer

Lens status: clouding of the lens Nuclear, Subcapsular and Cortical 0 - 0

1. - 1
2. - 2
3. - 3
4. - 4

Vitreous cells: number of cells per milimeter in the vitreous cavity 0 - 0 1 - traces 2 - +1 3 - +2 4 - +3 5 - +4

Vertical C/D ratio: relation between cup and optic nerve disc 0 - 0.1

1. - 0.2
2. - 0.3
3. - 0.4
4. - 0.5
5. - 0.6
6. - 0.7
7. - 0.8
8. - 0.9
9. - 1.0

Optic nerve edge: regularly over the optic disc 0 - Regular

1 - Irregular

Rim characteristic [ISNT pattern]: reduction pattern in the thickness of neural ring 0 - Conserved 1 - Not conserved

Peripapilar atrophy: presence of atrophy over the disc 0 - Alfa

1 - Beta 3 - Not apply

State of fovea: normality of the fovea 0 - normal

1 - abnormal

State of peripheral retina: state of the peripheral retina 0 - normal

1 - abnormal

State of choroid: choroidal health 0 - normal

1 - abnormal

After the visit 0, a 5 consecutive visits will be performed: for 1 day, 1 week, 1 month, 3 months and 6 months after the procedure. Identical data will be extracted, ophthalmological examination data, slit lamp exam, and the computerized visual fields (CVF) (CVF only at 3 and 6 months).

One member of the investigation team will collect all information during the follow-up time, and a second one member will review and collate data.

Statistical analysis will be performed in SPSS version 21. Univariate analyzes will perform; for categorical variables, frequency distribution will be made and reported in percentage, for the quantitative variables a measure of central tendency and dispersion will be made (mean, standard deviation and range) will calculate according to the relevance for each variable analyzed. Demographics such as age and gender variables will be described. For bivariate analysis comparing polytomous qualitative and quantitative variables (evolution of intraocular pressure with the type of trabeculoplasty used, number of antihypertensive medications required after the procedure with the type of trabeculoplasty, quantification of cellularity in the anterior chamber with type of trabeculoplasty) using parametric statistical analysis with ANOVA for independent samples and nonparametric with Kruskal-Wallis test. Also comparison of quantitative variables with quantitative variables (intraocular pressure before treatment and evolution of intraocular pressure after treatment) will be performed using the parametric inferential statistical Pearson correlation analysis and for nonparametric a Spearman correlation will be made. Finally, compare qualitative variables with qualitative variables (presence of peak intraocular pressure with type of laser trabeculoplasty performed) using the non-parametric statistical analysis Chi square test, Fisher exact test and Mac Nemar will make.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of either sex, aged ≥ 40 years
* Best distant visual acuity, better than or equal to 20/200
* Diagnosis of primary open-angle glaucoma, pseudoexfoliation glaucoma or pigmentary glaucoma, with open angles by Posner lens gonioscopy
* Intraocular pressure ≥ 20 mmHg, with medical treatment, as monotherapy or combination therapy.
* Previous computerized visual field within the six months previous performing trabeculoplasty
* Patients who understand and sign the informed consent
* Patient diagnosed with open-angle glaucoma who will undergo selective laser trabeculoplasty (SLT) with an amplitud of 360 degrees, or laser trabeculaplastia in pattern (PASCAL-Pattern Scan Laser) with an amplitud of 360 degrees. Made at initial session or in two 7 days separate sessions (each with session with an amplitude of180 degrees)

Exclusion Criteria:

* Advanced loss on visual field within 10 degrees of central fixation in a previous 3 months visual field
* Previous history of surgery for glaucoma management, except peripheral iridotomy
* Corneal disease that does not allow the use of applanation tonometer nor an accurate measurement of intraocular pressure
* Corneal disease which prevents adequate visualization of trabeculo by gonioscopy lens
* Use of topical or systemic steroids
* Concomitant participation in another study
* Coexistence of other ocular pathology different than cataract.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with Open-Angle Glaucoma with a non-optimal intraocular pressure control with topical/oral medications, who underwent to laser trabeculoplasty treatment, attending the Fundacion Oftalmológica Nacional between June 2014 and july 2016 on Bogotá-Colombia.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2014-09; Primary Completion 2016-09 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Intraocular pressure | Six months
  The eye pressure measured in millimeters of mercury, measure with Goldman tonometer at follow-up period

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Belalcazar, MD, Principal Investigator — Fundacion Oftalmológica Nacional
Locations (1):
- Fundacion Oftalmológica Nacional, Bogotá, Bogota D.C., Colombia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wang W, He M, Zhou M, Zhang X. Selective laser trabeculoplasty versus argon laser trabeculoplasty in patients with open-angle glaucoma: a systematic review and meta-analysis. PLoS One. 2013 Dec 19;8(12):e84270. doi: 10.1371/journal.pone.0084270. eCollection 2013. PMID 24367649
- [Background] Wise JB, Witter SL. Argon laser therapy for open-angle glaucoma. A pilot study. Arch Ophthalmol. 1979 Feb;97(2):319-22. doi: 10.1001/archopht.1979.01020010165017. No abstract available. PMID 575877
- [Background] Barkana Y, Belkin M. Selective laser trabeculoplasty. Surv Ophthalmol. 2007 Nov-Dec;52(6):634-54. doi: 10.1016/j.survophthal.2007.08.014. PMID 18029271
- [Background] Latina MA, Park C. Selective targeting of trabecular meshwork cells: in vitro studies of pulsed and CW laser interactions. Exp Eye Res. 1995 Apr;60(4):359-71. doi: 10.1016/s0014-4835(05)80093-4. PMID 7789416
- [Background] Sanghvi C, McLauchlan R, Delgado C, Young L, Charles SJ, Marcellino G, Stanga PE. Initial experience with the Pascal photocoagulator: a pilot study of 75 procedures. Br J Ophthalmol. 2008 Aug;92(8):1061-4. doi: 10.1136/bjo.2008.139568. Epub 2008 Jun 27. PMID 18586905
- [Background] Sambhara D, Aref AA. Glaucoma management: relative value and place in therapy of available drug treatments. Ther Adv Chronic Dis. 2014 Jan;5(1):30-43. doi: 10.1177/2040622313511286. PMID 24381726
- [Background] Buys YM. Economics of selective laser trabeculoplasty as primary therapy for glaucoma. Can J Ophthalmol. 2006 Aug;41(4):419-20. doi: 10.1016/S0008-4182(06)80001-3. No abstract available. PMID 16883356
- [Background] Quigley HA. Glaucoma. Lancet. 2011 Apr 16;377(9774):1367-77. doi: 10.1016/S0140-6736(10)61423-7. Epub 2011 Mar 30. PMID 21453963
- [Background] Samples JR, Singh K, Lin SC, Francis BA, Hodapp E, Jampel HD, Smith SD. Laser trabeculoplasty for open-angle glaucoma: a report by the american academy of ophthalmology. Ophthalmology. 2011 Nov;118(11):2296-302. doi: 10.1016/j.ophtha.2011.04.037. Epub 2011 Aug 17. PMID 21849211
- [Background] Krasnov MM. [Laser puncture of the anterior chamber angle in glaucoma (a preliminary report)]. Vestn Oftalmol. 1972;3:27-31. No abstract available. Russian. PMID 5078295
- [Background] Van Buskirk EM, Pond V, Rosenquist RC, Acott TS. Argon laser trabeculoplasty. Studies of mechanism of action. Ophthalmology. 1984 Sep;91(9):1005-10. doi: 10.1016/s0161-6420(84)34197-5. PMID 6493712
- [Background] Alvarado JA, Alvarado RG, Yeh RF, Franse-Carman L, Marcellino GR, Brownstein MJ. A new insight into the cellular regulation of aqueous outflow: how trabecular meshwork endothelial cells drive a mechanism that regulates the permeability of Schlemm's canal endothelial cells. Br J Ophthalmol. 2005 Nov;89(11):1500-5. doi: 10.1136/bjo.2005.081307. PMID 16234461
- [Background] Bradley JM, Anderssohn AM, Colvis CM, Parshley DE, Zhu XH, Ruddat MS, Samples JR, Acott TS. Mediation of laser trabeculoplasty-induced matrix metalloproteinase expression by IL-1beta and TNFalpha. Invest Ophthalmol Vis Sci. 2000 Feb;41(2):422-30. PMID 10670472
- [Background] The Glaucoma Laser Trial (GLT). 2. Results of argon laser trabeculoplasty versus topical medicines. The Glaucoma Laser Trial Research Group. Ophthalmology. 1990 Nov;97(11):1403-13. PMID 2255512
- [Background] Bylsma SS, Samples JR, Acott TS, Van Buskirk EM. Trabecular cell division after argon laser trabeculoplasty. Arch Ophthalmol. 1988 Apr;106(4):544-7. doi: 10.1001/archopht.1988.01060130590044. PMID 3355425
- [Background] Pham H, Mansberger S, Brandt JD, Damji K, Ramulu PY, Parrish RK. Argon laser trabeculoplasty versus selective laser trabeculoplasty. Surv Ophthalmol. 2008 Nov-Dec;53(6):641-6. doi: 10.1016/j.survophthal.2008.08.020. PMID 19026324
- [Background] Zhao JC, Grosskreutz CL, Pasquale LR. Argon versus selective laser trabeculoplasty in the treatment of open angle glaucoma. Int Ophthalmol Clin. 2005 Fall;45(4):97-106. doi: 10.1097/01.iio.0000176370.01511.6e. No abstract available. PMID 16199969
- [Background] Wang H, Cheng JW, Wei RL, Cai JP, Li Y, Ma XY. Meta-analysis of selective laser trabeculoplasty with argon laser trabeculoplasty in the treatment of open-angle glaucoma. Can J Ophthalmol. 2013 Jun;48(3):186-92. doi: 10.1016/j.jcjo.2013.01.001. PMID 23769780
- See also: Selective laser trabeculoplasty versus argon laser trabeculoplasty in patients with open-angle glaucoma: a systematic review and meta-analysis — http://www.ncbi.nlm.nih.gov/pubmed/24367649
- See also: Argon laser therapy for open-angle glaucoma. A pilot study — http://www.ncbi.nlm.nih.gov/pubmed/575877
- See also: Selective laser trabeculoplasty — http://www.ncbi.nlm.nih.gov/pubmed/18029271
- See also: Selective targeting of trabecular meshwork cells: in vitro studies of pulsed and CW laser interactions — http://www.ncbi.nlm.nih.gov/pubmed/7789416
- See also: Initial experience with the Pascal photocoagulator: a pilot study of 75 procedures — http://www.ncbi.nlm.nih.gov/pubmed/18586905
- See also: Glaucoma management: relative value and place in therapy of available drug treatments — http://www.ncbi.nlm.nih.gov/pubmed/24381726
- See also: Economics of selective laser trabeculoplasty as primary therapy for glaucoma — http://www.ncbi.nlm.nih.gov/pubmed/16883356
- See also: Glaucoma — http://www.ncbi.nlm.nih.gov/pubmed/21453963
- See also: Laser trabeculoplasty for open-angle glaucoma: a report by the american academy of ophthalmology — http://www.ncbi.nlm.nih.gov/pubmed/21849211
- See also: Laser puncture of the anterior chamber angle in glaucoma (a preliminary report) — http://www.ncbi.nlm.nih.gov/pubmed/5078295
- See also: Argon laser trabeculoplasty. Studies of mechanism of action — http://www.ncbi.nlm.nih.gov/pubmed/6493712
- See also: A new insight into the cellular regulation of aqueous outflow: how trabecular meshwork endothelial cells drive a mechanism that regulates the permeability of Schlemm's canal endothelial cells — http://www.ncbi.nlm.nih.gov/pubmed/16234461
- See also: Mediation of laser trabeculoplasty-induced matrix metalloproteinase expression by IL-1beta and TNFalph — http://www.ncbi.nlm.nih.gov/pubmed/10670472
- See also: Results of argon laser trabeculoplasty versus topical medicines. The Glaucoma Laser Trial Research Group — http://www.ncbi.nlm.nih.gov/pubmed/2255512
- See also: Trabecular cell division after argon laser trabeculoplasty — http://www.ncbi.nlm.nih.gov/pubmed/3355425
- See also: Argon laser trabeculoplasty versus selective laser trabeculoplasty — http://www.ncbi.nlm.nih.gov/pubmed/19026324
- See also: Argon versus selective laser trabeculoplasty in the treatment of open angle glaucom — http://www.ncbi.nlm.nih.gov/pubmed/16199969
- See also: Meta-analysis of selective laser trabeculoplasty with argon laser trabeculoplasty in the treatment of open-angle glaucoma — http://www.ncbi.nlm.nih.gov/pubmed/23769780